CLINICAL TRIAL: NCT05737602
Title: Promoting Stress Management and Resilience Among Individuals With Von Hippel- Lindau Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Rappaport Foundation (Unknown); The Claflin Distinguished Scholar Awards (Unknown)
Responsible Party: Principal Investigator, Giselle K. Perez Lougee, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-612
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Von Hippel-Lindau Disease; Genetic Disorder
Keywords: Von-Hippel-Lindau Disease; VHL; Genetic Disorder
MeSH Terms: conditions — von Hippel-Lindau Disease; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3RP-VHL (Experimental): * An adapted version of the 3RP (3RP-VHL) for individuals with VHL. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies. It will be delivered in weekly sessions over the course of approximately 8 weeks.
  * Complete pre- and post-intervention surveys.
  Interventions: Behavioral: 3RP-VHL

INTERVENTIONS:
Behavioral: 3RP-VHL — An adapted version of the Relaxation Response Resiliency Program (3RP) for individuals with VHL.
  Other Names: Relaxation Response Resiliency Program for VHL

SUMMARY:
The Relaxation Response Resiliency Program (3RP) has shown efficacy in improving coping and resilience across diverse populations; however, little is known about how it helps individuals manage the challenges of living with a chronic illness. This study proposes to pilot test an adapted version of the 3RP among patients living with VHL.

DETAILED DESCRIPTION:
The 3RP has not been carried out with VHL patients. As such, the investigators are looking to see if an adapted program, tailored to the needs of patients with VHL, is feasible, acceptable, and helpful in improving coping among individuals living with VHL.

This study is a two phase trial. Phase I is descriptive. It is comprised of conducting interviews with patients and caregivers to understand the challenges of living with VHL and patient's programatic needs. This information will be used to tailor the program for patients living with VHL. Phase II is a single-arm feasibility trial that will examine if the adapted program is feasible, acceptable, and helps promote stress management among VHL patients. To these means, we will test the adapted 3RP (3RP-VHL) in up to 40 patients living with VHL. Participants will complete surveys at baseline and post 3RP-VHL program completion. This record will reflect the trial component (Phase II) only, as feasibility and acceptability outcomes will be collected for this phase.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18+
* Confirmed diagnosis of VHL

Exclusion Criteria:

* Is medically, psychiatrically, or otherwise unable to participate (as determined by a physician or study PI).
* Unwilling or unable to participate in study sessions delivered via Partners Telehealth videoconferencing.
* Participated in Phase 1 qualitative interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
3RP-VHL Feasibility: Percent of Identified Eligibles Who Enroll | Post-treatment completion (treatment is approximately 2 months)
  Percent of identified eligibles who were approached (hence given the opportunity to participate) who enroll (i.e., sign consent and complete baseline).
3RP-VHL Feasibility: Proportion of Participants Completing the 3RP-VHL Program | Post-treatment completion (treatment is approximately 2 months)
  Among those who initiated the program, this is the proportion of patients who completed the program (defined as completing 6 out of 8 sessions). Participants who complete at least 75% of the treatment sessions (6 out of 8 sessions) will be identified as treatment completers.
3RP-VHL Acceptability: Five Questions | Post-treatment completion (treatment is approximately 2 months)
  Acceptability will be assessed with five questions rated on a 4-point Likert scale (1=not at all to 4=very). More specifically, acceptability will be defined as ≥75% of responses rated at least 3/4 on enjoyableness, convenience, helpfulness, future use, and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Perez, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu